CLINICAL TRIAL: NCT00430768
Title: Preclinical & Phase I/II Trials of AAV-AAT Vectors: Phase I Trial of Intramuscular Injection of a Recombinant Adeno-Associated Virus Alpha 1-Antitrypsin (rAAV1-CB-hAAT) Gene Vector to AAT-Deficient Adults
Brief Title: Experimental Gene Transfer Procedure to Treat Alpha 1-Antitrypsin (AAT) Deficiency
Acronym: AAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Beacon Therapeutics (Industry); Alpha-1 Foundation (Other); University of Florida (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Terence Flotte, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 438; 5R01HL069877 (NIH); NIH-OBA 0404-638 (Registry Identifier: Gene Therapy Protocol Number); NCRR-supported GCRC# 611 (Other: University of Florida); UF IBC RD 2630 (Other: University of Florida); AGTC-AAV1-001 (Other: Applied Genetics Technologies C); WIRB # 20052374 (Other: Western Institutional Review B); BB-IND 12728 (Other: FDA); RR00032, RR00082 (Other Grant/Funding Number: NCRR)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Gene Transfer Techniques; Gene Therapy; AAV; AAT; Phase I; Intramuscular transfer
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 Low Dose (Experimental): rAAV1-CB-hAAT 6.9 x10e12 vector genomes (vg) administered in a 9.9 ml volume of study agent in nine separate 1.1 mL injections in the deltoid muscle of the "non-dominant" side under ultrasound guidance
  Interventions: Biological: rAAV1-CB-hAAT
- Group 2 Middle Dose (Experimental): rAAV1-CB-hAAT 2.2 x 10e13 vg administered in a 9.9 ml volume of study agent in nine separate 1.1 mL injections in the deltoid muscle of the "non-dominant" side under ultrasound guidance
  Interventions: Biological: rAAV1-CB-hAAT
- Group 3 High Dose (Experimental): rAAV1-CB-hAAT 6.0 x10e13 vg administered in a 9.9 ml volume of study agent in nine separate 1.1 mL injections in the deltoid muscle of the "non-dominant" side under ultrasound guidance
  Interventions: Biological: rAAV1-CB-hAAT

INTERVENTIONS:
Biological: rAAV1-CB-hAAT

SUMMARY:
Individuals with a deficiency of the alpha 1-antitrypsin (AAT) protein are at risk for developing emphysema and liver damage. Researchers have developed a way to introduce normal AAT genes into muscle cells with the expectation that the AAT protein may be produced at normal levels. This study will evaluate the safety of the experimental gene transfer procedure in individuals with AAT deficiency. The study will also determine what dose may be required to achieve normal levels of AAT.

DETAILED DESCRIPTION:
AAT deficiency is a genetic disorder in which individuals have inadequate levels of the AAT protein. AAT protects the lungs from white blood cell enzymes that can damage air sacs within the lungs, potentially leading to emphysema. Experimental gene transfer procedures, in which normal copies of genes are inserted into cells, are being developed to treat many genetic diseases, including AAT deficiency. In this study, a modified virus, adeno-associated virus (AAV), has been genetically engineered to contain a normal copy of the AAT gene. When AAV is combined with the AAT gene, the resulting agent, Recombinant Adeno-Associated Virus Alpha 1-Antitrypsin (rAAV1-CB-hAAT) Gene Vector with a chicken beta actin promoter (CB), may be able to carry normal copies of the AAT gene into muscle cells with the expectation that additional AAT would be produced. The purpose of this study is to evaluate the safety of injecting rAAV1-CB-hAAT into individuals with AAT deficiency.

This 14-month study will enroll individuals with AAT deficiency. Participants currently using AAT protein replacement will discontinue its use for 19 weeks during the study. Participants will first attend a baseline study visit, which will include a medical history review; a physical examination; an electrocardiogram (ECG) to record heart activity; blood, urine, and semen collection; pulmonary function tests; and chest and arm scans. Participants will then attend a 5-day inpatient visit, during which they will receive a series of injections consisting of one of four different doses of rAAV1-CB-hAAT. Physical examinations will occur on all 5 inpatient days; pulmonary function testing, arm circumference measurements, and collection of blood, urine, and semen will occur on selected days of the inpatient stay. Follow-up study visits, with possible overnight stays, will occur on Days 14 and 90. On Days 30, 45, 60, 75, 180, 270, and 365, participants will have blood drawn at a local clinic. On these same days, study staff will contact participants by telephone to review their medical history and symptoms. Unused blood and semen samples will be frozen and stored for future research purposes. Participants will have yearly follow-up evaluations by either telephone or mail for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AAT deficiency
* Forced expiratory volume in one second (FEV1) greater than 24% of predicted value (post bronchodilator)
* Willing to discontinue AAT protein replacement 4 weeks (Group 1) and 8 weeks (Groups 2 and 3) prior to study entry, and to resume 11 weeks after rAAV1-CB-hAAT has been administered
* Willing to discontinue aspirin, aspirin-containing products, and other drugs that may alter platelet function 7 days prior to study entry, and to resume 24 hours after rAAV1-CB-hAAT has been administered
* Willing to use contraception throughout the study

Exclusion Criteria:

* Required antibiotic therapy for a respiratory infection in the 28 days prior to rAAV1-CB-hAAT administration
* Required oral or systemic corticosteroids in the 28 days prior to rAAV1-CB-hAAT administration
* Liver disease
* Currently receiving or has received an investigational study agent in the 30 days prior to study entry
* Received gene transfer agents in the 6 months prior to study entry
* Currently smokes cigarettes or uses illegal drugs
* History of immune response to human AAT replacement
* History of platelet dysfunction
* Abnormal ECG, heart disease, pulmonary edema, or embolism in the 6 months prior to study entry
* Current or recent facial or chest trauma that makes it medically impossible to perform pulmonary function tests (PFTs)
* Any other medical condition that the investigator deems unsuitable for study participation
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence R. Flotte, MD, Principal Investigator — UMass Medical School; Mark L Brantly, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, College of Medicine, Department of Pediatrics, Gainesville, Florida
  - University of Massachusetts School of Medicine, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Laboratory information shared as received; copy of manuscript given to patients; at 5 year follow up Principal investigator explained results to patients

REFERENCES:
- [Background] Song S, Morgan M, Ellis T, Poirier A, Chesnut K, Wang J, Brantly M, Muzyczka N, Byrne BJ, Atkinson M, Flotte TR. Sustained secretion of human alpha-1-antitrypsin from murine muscle transduced with adeno-associated virus vectors. Proc Natl Acad Sci U S A. 1998 Nov 24;95(24):14384-8. doi: 10.1073/pnas.95.24.14384. PMID 9826709
- [Background] Lu Y, Choi YK, Campbell-Thompson M, Li C, Tang Q, Crawford JM, Flotte TR, Song S. Therapeutic level of functional human alpha 1 antitrypsin (hAAT) secreted from murine muscle transduced by adeno-associated virus (rAAV1) vector. J Gene Med. 2006 Jun;8(6):730-5. doi: 10.1002/jgm.896. PMID 16518879
- [Background] Brantly ML, Spencer LT, Humphries M, Conlon TJ, Spencer CT, Poirier A, Garlington W, Baker D, Song S, Berns KI, Muzyczka N, Snyder RO, Byrne BJ, Flotte TR. Phase I trial of intramuscular injection of a recombinant adeno-associated virus serotype 2 alphal-antitrypsin (AAT) vector in AAT-deficient adults. Hum Gene Ther. 2006 Dec;17(12):1177-86. doi: 10.1089/hum.2006.17.1177. PMID 17115945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited to the University of Florida, Clinical Research Center for the active study; long term follow up was completed at the University of Massachusetts, Medical School.
Pre-assignment Details: Subjects on alpha-1 antitrypsin (AAT) protein replacement product prior to study, discontinued treatment 4 weeks (Group 1) and 8 weeks (Groups 2 and 3) prior to study agent administration and were able to resume treatment 11 weeks after study agent had been administered. The group was determined by when the subject joined the study.
Groups:
- Group 1 Low Dose: 6.9 x10e12 vector genomes (vg)
  Group 1 receives rAAV1-CB-hAAT 6.9 x10e12 vg.
- Group 2 Middle Dose: 2.1 x 10e13 vector genomes; 2.2 x 10e13 vector genomes
  Group 2, 1 subject received rAAV1-CB-hAAT 2.1 x10e13 vg; 202 and 203 received rAAV1-CB-hAAT 2.2 x10e13 vg
- Group 3 High Dose: rAAV1-CB-hAAT 6.0 x10e13 vg
  Group 3 receives rAAV1-CB-hAAT 6.0 x10e13 vg
Period: Overall Study
Arm/Group | Group 1 Low Dose | Group 2 Middle Dose | Group 3 High Dose
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Low Dose: 6.9 x10e12 vector genomes
  Group 1 receives rAAV1-CB-hAAT 6.9 x1012 vg (vector genomes), e
- Group 2 Middle Dose: 2.1 x 10e13 vector genomes
  Group 2 receives rAAV1-CB-hAAT 2.1 x1013 vg
- Group 3 High Dose: rAAV1-CB-hAAT 6.0 x10e13 vg
  Group 2 receives rAAV1-CB-hAAT 2.1 x1013 vg
- Total: Total of all reporting groups
Arm/Group | Group 1 Low Dose | Group 2 Middle Dose | Group 3 High Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Customized [Median (Full Range); unit: years] | 69 [66 to 73] | 54 [38 to 59] | 47 [35 to 61] | 54 [35 to 73]
Gender [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 4
  Male | 1 | 3 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9
FEV1 (% predicted) [Median (Full Range); unit: percent predicted] — forced expiratory volume in 1 second; percent predicted for race, height, and weight
  percent predicted | 86.7 [53.6 to 92.1] | 50.8 [40.5 to 93.0] | 58.0 [54.9 to 97.6] | 58.0 [40.5 to 97.6]
Weight (kg) [Median (Full Range); unit: kilograms] | 66.5 [54.6 to 73.7] | 83.0 [72.7 to 89.0] | 72.6 [69.3 to 134.6] | 72.6 [54.6 to 134.6]
Prior AAT Protein Augmentation Therapy [Number; unit: participants]
  Yes | 2 | 1 | 1 | 4
  No | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Possibly, Probably or Definitely Related to Study Drug
Description: Adverse events considered possibly, probably or definitely related to study drug/study drug procedure Criteria to evaluate severity according to Attachment 2 of the Protocol
  1. Mild toxicity, usually transient, requiring no special treatment and generally not interfering with usual daily activities
  2. Moderate toxicity which may be ameliorated by simple therapeutic maneuvers, and impairs usual activities
  3. Severe toxicity which requires therapeutic intervention and interrupts usual activities. Hospitalization may or may not be required
  4. Life-threatening toxicity which requires hospitalization
Time Frame: During 1 year after study agent administration
Population: subjects in the group reporting the event
Measure: Number; unit: participants
Arm/Group | Group 1 Low Dose | Group 2 Middle Dose | Group 3 High Dose
Number analyzed (Participants) | 3 | 3 | 3
participants
  Number with one or more related AE | 2 | 2 | 3
  injection site erythema mild | 2 | 0 | 0
  Inject site hematoma mild | 1 | 2 | 3
  Inject site induration mild | 1 | 0 | 0
  Inject site pain mild | 0 | 0 | 1
  Inject site swelling mild | 1 | 1 | 0
  Injection site warmth | 0 | 1 | 0

2. Secondary Outcome: hAAT Expression in Blood Measured Using M-specific Allele ELISA
Description: 4 subjects received prior AAT augmentation therapy; 2 subjects from Group 1 having only washed out for only 28 days complicated the measurement of M-specific levels 2 subjects from group 1 and the other subject did not have an appreciable change in M-specific AAT levels. Thus reporting only Cohorts 2 and 3. After day 90 patients were able to resume AAT protein therapy and thus levels were not collected following commencement of therapy on 201 and 303. 202, Day 365 blood hemolyzed; level not determinable.
Time Frame: Baseline, Days 14, 30, 45, 60, 90, (180, 270, and 365 if not on protein replacement therapy)
Population: AAT Levels of each subject at various time points Baseline and Days following administration. 202 Day 365 blood hemolyzed; not determinable, 201 and 303 went back on AAT protein augmentation therapy after day 90, unable to collect M-specific levels on day 180, 270 and 303.
Measure: Number; unit: nM
Groups:
- 201 (Medium Dose): Subject 201 M-specific AAT Level
- 202 (Medium Dose): Subject 202 M-specific AAT Level
- 203 (Medium Dose): Subject 203 M-specific AAT Level
- 301 (High Dose): Subject 301M-specific AAT Level
- 302 (High Dose): Subject 302 M-specific AAT Level
- 303 (High Dose): Subject 303 M-specific AAT Level
Arm/Group | 201 (Medium Dose) | 202 (Medium Dose) | 203 (Medium Dose) | 301 (High Dose) | 302 (High Dose) | 303 (High Dose)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
nM
  Baseline Level | 33 | 10.8 | 11.2 | 9.6 | 7.1 | 18.3
  Day 14 Level | 7.5 | 12.7 | 12.0 | 13.2 | 10.3 | 7.8
  Day 30 Level | 7.5 | 17.8 | 14.7 | 24.7 | 16.6 | 10.5
  Day 45 Level | 6.2 | 16.7 | 14.5 | 22.6 | 18.5 | 41.5
  Day 60 Level | 15.1 | 16.8 | 20.7 | 20.8 | 10.5 | 37.7
  Day 75 Level | 14.6 | 14.7 | 12.9 | 21.8 | 14.3 | 45.9
  Day 90 Level | 26.8 | 12.6 | 14.6 | 42.6 | 6.7 | 48.5
  Day 180 Level | NA — resumed AAT protein therapy | 9.8 | 10.8 | 41.7 | 26.4 | NA — resumed AAT protein therapy
  Day 270 Level | NA — resumed AAT protein therapy | 8.0 | 7.0 | 47.9 | 33.5 | NA — resumed AAT protein therapy
  Day 365 Level | NA — resumed AAT protein therapy | NA — blood hemolyzed | 24.2 | 50.9 | 33.4 | NA — resumed AAT protein therapy

ADVERSE EVENTS:
Time Frame: 1 year active study; 4 years long term follow up
Groups:
- Group 1 Low Dose: 6.9 x10e12 vector genomes
  e. Group 1 receives rAAV1-CB-hAAT 6.9 x10e12 vg (vector genomes)
- Group 2 Middle Dose: 2.2 x 10e13 vector genomes
  Group 2 receives rAAV1-CB-hAAT 2.1 x10e13 vg
Arm/Group | Group 1 Low Dose | Group 2 Middle Dose | Group 3 High Dose
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Low Dose (N=3) | Group 2 Middle Dose (N=3) | Group 3 High Dose (N=3)
E. coli Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — 69 y/o man low dose of study drug 14MAR2006. 6 Apr 2006 diagnosed with E coli epididymitis confirmed by testicular ultrasound and urine culture. Event considered not related to study agent.
Pharyngoesophageal diverticulum repair with complications (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Subject received study agent 14Mar2006.Surgical repair 20Jan2010 for pharyngoesophageal diverticulum.Hospitalized 27Jan2010 with GI anastomotic leak following surgery, treated with feeding tube, resolved, considered not related to study agent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Low Dose (N=3) | Group 2 Middle Dose (N=3) | Group 3 High Dose (N=3)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site hematoma (General disorders) | 1 (1) | 2 (2) | 3 (3)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyl transferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Long Term Follow up
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Long Term Follow up
Prostate Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Long Term Follow up
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Long Term Follow up

LIMITATIONS AND CAVEATS:
Study results based on small number of subjects No statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less